CLINICAL TRIAL: NCT01720407
Title: Relevance of Imiquimod as Neo-adjuvant Treatment to Reduce Excision Size and the Risk of Intralesional Excision in Lentigo Malignant of the Face
Acronym: ImiReduc
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: MEDA Pharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD/11/06-S
Record Dates: First submitted 2012-10-23; First posted 2012-11-02 (Estimated); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Lentigo Maligna Melanoma (Head or Neck)
Keywords: Dermatology/ Skin cancers/Lentigo maligna melanoma
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Masking Description: Surgeon does not know the result of randomization.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imiquimod (Experimental)
  Interventions: Drug: Imiquimod cream + surgery
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo + surgery

INTERVENTIONS:
Drug: Imiquimod cream + surgery — Imiquimod (5 times per week) applied to and extending 1cm beyond the lesion for a period of 4 weeks (i.e. a total of 20 applications), followed by surgery performed four weeks after the last application of the topical treatment. If excision is intralesional, re-excision at 5mm will be performed within a few days (equivalent to 2-stage surgery).
  Arms: Imiquimod
Drug: Placebo + surgery — Placebo (5 times per week) applied to and extending 1cm beyond the lesion for a period of 4 weeks, followed by surgery performed four weeks after the last application of the topical treatment. If excision is intralesional, re-excision of 5mm of clinically healthy tissue will be performed within a few days (equivalent to 2-stage surgery).
  Arms: Placebo

SUMMARY:
Lentigo malignant (LM) is an intraepidermal melanocytic proliferation occurring on photoexposed skin. In our project, this term applies both to Dubreuilh's melanosis and to Dubreuilh's intraepidermal melanoma. It consequently excludes invasive melanoma. Although surgery is the treatment of choice, it remains without consensus on the margins (5 mm or 10 mm) excision for a localized tumor on the face.

Several studies have shown that imiquimod, activating local immunity by interferon production, induced LM or MLM regression and could also decrease the frequency of relapses.

The principal aim of our project is to study the effect of imiquimod versus placebo in pre-operative neoadjuvant treatment aimed at reducing both surgical margins, as from the first surgical procedure, and the frequency of short and medium term recurrence of LM. Furthermore, the improvement in patient quality of life could also be significant.

DETAILED DESCRIPTION:
The primary endpoint of the study is to demonstrate that neoadjuvant treatment of LM by imiquimod prior to surgery can reduce the frequency of intralesional excisions as from the first surgical procedure, with a healthy tissue margin of 5mm. Furthermore, the improvement in patient quality of life could also be significant.

The number of patients to be included in the study is 268.

For each patient, the study will involve several stages (S), as follows:

S0 (Selection): information and obtaining of the patient's informed consent. Performance of biopsy for histological confirmation of LM

S1 (S0 + ~ 2 weeks): patient inclusion following anatomopathological confirmation of LM. Patient randomisation in one or other study arm: imiquimod versus placebo and initiation of topical treatment.

S2 (S1 + 4 weeks): Discontinuation of imiquimod/placebo application. Scheduling of the surgical procedure 4 weeks later.

S3 (S2 + 4 weeks): Surgery.

S4: After the last surgical procedure, simple clinical follow up will be ensured every 6 months for a period of 3 years, in order to study the recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients from both sexes aged over 18 years and operable
* Presenting with LM of the face, the neck, or the scalp (in case of hairless scalp only) histologically confirmed by biopsy
* Patients presenting with a primitive lesion, of a surface ≥ to 1cm² and ≤ to 20cm², with the possibility of graft or flap reconstruction
* LM previously untreated by surgery
* LM without prior treatment with liquid nitrogen or any other local treatment within 3 months
* ECOG ≤ 2
* Leucocytes ≥ 3,000/mm³
* Neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Haemoglobin ≥ 9.0g/dL
* Absence of severe evolutive infection
* Absence of known HIV infection
* Absence of corticotherapy and treatment by immunosuppressive agents
* Absence of excoriation and scarring biopsy prior to application of study treatment
* Membership to a social security insurance scheme.
* Negative pregnancy test conducted during the inclusion consultation for non-menopausal women.
* Effective contraception for patients of childbearing age
* Signed informed consent

Exclusion Criteria:

* LM located on the eyelids are excluded, together with LM in anatomic sites other than the face, the neck or the scalp
* Melanomas other than LM
* Invasive LM
* LM with a surface area < to 1cm² or > to 20cm²
* LM of which the macroscopic contours cannot be defined
* Patients who are allergic to imiquimod excipient (eg hydroxybenzoate)
* Patients with a hypersensitivity to active substances or to any of the excipients of the placebo (for example propyl parahydroxybenzoate)
* Patients treated by immunosuppressive agents, immunomodulators, cytotoxic agents or corticosteroids (local and systemic) during the 4-week period prior to the selection visit
* Patients with auto-immune disease (except vitiligo) or transplant patients
* Cutaneous reconstruction not possible
* Presence of associated evolutive neoplasia since less than 5 years (with the exception of basal cell carcinoma, Bowen's carcinoma and carcinoma in situ of the cervix)
* Patient refusing surgery under local or general anaesthesia
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the margin of resection. Success is defined by an extralesional excision as from the first surgical procedure performed with a healthy tissue margin of 5 mm. | 10 weeks

SECONDARY OUTCOMES:
The number of surgical re-excisions required to obtain complete remission. | Baseline, 2 months till 3 years
The number of recurrences, defined as the reappearance of pigmentation within 3 years of surgical excision. | Baseline, 2 months till 3 years
The number of histologically confirmed complete remissions under imiquimod. | Baseline, 2 months till 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Dréno, MD, PhD, Principal Investigator — Nantes University Hospital
Locations (22):
- France (22):
  - CHU, Besançon
  - CHU Hôpital Haut-Lévêque, Bordeaux
  - CHU Hôpital Saint André, Bordeaux
  - AP-HP Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHU, Brest
  - CHU Michallon, Grenoble
  - CH, Le Mans
  - CHRU, Lille
  - CHU, Limoges
  - CHU, Lyon
  - AP-HM, Marseille
  - CHU, Montpellier
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - CHU, Nice
  - CHU, Orléans
  - AP-HP Hôpital Saint Louis, Paris
  - CHU Milétrie, Poitiers
  - CHU, Reims
  - CHU Pontchaillou, Rennes
  - CHU, Saint-Etienne
  - Chu (Iucto), Toulouse
  - CHU, Tours

REFERENCES:
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215